CLINICAL TRIAL: NCT01476280
Title: A Randomized Double Blind Study to Evaluate Efficacy of Ramosetron and Palonosetron for Prevention of Postoperative Nausea and Vomiting After Gynaecological Laparoscopic Surgery
Brief Title: Palonosetron Versus Ramosetron for the Prevention of Postoperative Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Incheon St.Mary's Hospital (Other)
Responsible Party: Principal Investigator, Soo Kyoung Park, Clinical professor, Incheon St.Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OC11MISI0027
Record Dates: First submitted 2011-11-15; First posted 2011-11-22 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: antiemetics; ramosetron; palonosetron; PONV(postoperative nausea and vomiting)
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Palonosetron; ramosetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Palonosetron (Sham Comparator)
  Interventions: Drug: palonosetron
- Ramosetron (Sham Comparator)
  Interventions: Drug: Ramosetron

INTERVENTIONS:
Drug: palonosetron — 0.075mg immediately before induction of anesthesia
  Arms: Palonosetron
Drug: Ramosetron — 0.3mg immediately before induction of anesthesia
  Arms: Ramosetron

SUMMARY:
Ramosetron and palonosetron are more recently developed 5-hydroxytryptamine type 3 receptor antagonists and this randomized double blind study was designed to compare efficacy of ramosetron and palonosetron to prevent postoperative nausea and vomiting. Investigator hypothesized that palonosetron would have stronger and longer lasting antiemetic effect compared with ramosetron and evaluated the patients for the first 48 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA Physical Status 1 or 2
* Elective gynaecological laparoscopic surgery of ≥ 1h duration

Exclusion Criteria:

* Anti-emetics, steroids, or psychoactive medications within 24 h of study initiation
* Vomiting or retching in the 24 h preceding surgery
* Cancer chemotherapy within 4 weeks or emetogenic radiotherapy within 8 weeks before study entry
* Ongoing vomiting from gastrointestinal disease

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative nausea and vomiting for 48 hours after surgery | for 48 hours after surgery

SECONDARY OUTCOMES:
severity of nausea for 48 hours after surgery | for 48 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Soo Kyoung Park, Principal Investigator — Incheon St.Mary's Hospital
Locations (1):
- Incheon St. Mary's hospital, Incheon, South Korea